CLINICAL TRIAL: NCT06150456
Title: Evaluation of Alveolar Bone Preservation After Molar Extraction Using Photobiomodulation Combined With Grafting With Scaffold Biomaterial: Clinical, Randomized, Triple-blind Study.
Brief Title: Study of Alveolar Bone Preservation Using Photobiomodulation Combined With Grafting With Scaffold Biomaterial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, PHD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vanessa 1
Record Dates: First submitted 2023-11-09; First posted 2023-11-29 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Extracting Own Teeth; Bone Substitutes
Keywords: Bone regeneration; photobiomodulation; scaffold biomaterial
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental: Group 1 (Experimental): 15 patients who will only have their first teeth or second molars extracted.
  Interventions: Procedure: extraction
- Experimental: Group 2 (Experimental): 15 patients who will have only their first or second molars extracted and will receive infrared laser treatment
  Interventions: Procedure: extraction; Radiation: low level laser therapy
- Experimental: Group 3 (Experimental): 15 patients who will have their first or second molars extracted and will receive a graft with scaffold biomaterial
  Interventions: Procedure: extraction; Biological: Plenum® OSShp and Plenum® Guide
- Experimental: Group 4 (Experimental): 15 patients who will have their first or second molars extracted and will receive a graft with scaffold biomaterial and infrared laser treatment
  Interventions: Procedure: extraction; Radiation: low level laser therapy; Biological: Plenum® OSShp and Plenum® Guide

INTERVENTIONS:
Procedure: extraction — extraction: in all groups, extraction will be performed
Radiation: low level laser therapy — extraction: in all groups, extraction will be performed Treatment with low-intensity infrared 808 nm laser therapy will be applied in 2 stages: one in the immediate postoperative period and 10 days after surgery.
  Arms: Experimental: Group 2; Experimental: Group 4
Biological: Plenum® OSShp and Plenum® Guide — extraction: in all groups, extraction will be performed Immediately after tooth extraction, the biomaterials Plenum® OSShp and Plenum® Guide (Brazil) will be added to the dental socket, serving as a bone substitute and maintaining alveolar dimensions.
  Arms: Experimental: Group 3; Experimental: Group 4

SUMMARY:
Bone graft added to the dental socket immediately after tooth extraction prevents atrophy and deformity of the bone at the site of element loss, enabling rehabilitation with implants. Photobiomodulation accelerates bone healing; stimulates blood flow; activates osteoblasts, decreases osteoclastic activity, and improves the integration of the biomaterial with bone tissue. The study aims to develop a protocol for the management and preservation of alveolar bone after the loss of first and/or second permanent molars in patients aged between 8 and 17 years, with an indication for extraction associated or not with 808 nm infrared laser treatment. . Materials and methods: 60 patients aged between 8 and 17 years will be randomized and randomly divided into 4 groups, n= 15: Exo (extraction), Exo+Laser (extraction and laser treatment), Exo+Biomat (extraction with graft biomaterial), Exo+Biomat+Laser (biomaterial extraction and grafting and laser treatment). The biomaterials of choice will be Plenum® OSShp and Plenum® Guide (Brazil), added to the alveolus immediately after molar extraction, groups that will receive the laser (λ = 808 nm, power = 100 mW, radiant energy 3J per point in 3 buccal, occlusal and lingual/palatal points), will receive the irradiation in the surgical act, 48 hours and 10 days after the surgery, in the Exo and Exo+Biomat groups a similar laser device without emission of irradiation will be used, the operator who will apply the laser and the patient will be blind to the device used and the patient will not know whether or not he received the biomaterial. Analysis: computed tomography and intraoral scanning were performed pre-surgery, 3 and 6 months after surgery; to assess bone volume by measuring the height and width of the socket in each group, as well as trabecular bone and the interdental space of the teeth lateral to the missing element. Statistical analysis will be performed using the Shapiro-Wilks test, Student's t-test, or Wilcoxon-Mann-Whitney test for parametric and non-parametric data, respectively, they will be two-tailed and the significance level adopted will be α = 0.05.

DETAILED DESCRIPTION:
Clinical, randomized, triple-blind, triple-blind study (the patient will not know whether or not he has received the laser treatment or grafted with the biomaterial, and the operator who will apply the laser will also be blinded to the device with or without laser irradiation.

60 participants will be recruited to attend the dentistry clinic of Universidade Nove de Julho, in the courses of surgery, endodontics, and pediatric dentistry, as well as in a private office, with an indication for the removal of first and second upper and lower molars. This recruitment will only take place after approval by the ethics committee.

4.3 Sample size: The sample size was determined based on the primary outcome of the study: alveolar preservation with scaffold biomaterial. Based on data from Rosero et al. (Photobiomodulation as adjuvant therapy for alveolar preservation: a preliminary study in humans) and Araújo et al. (Ridge changes after engraftment of fresh extraction sockets in man. A randomized clinical trial) Our initial sample size estimate was 9 subjects per group for a significant level of 0.05 and an estimated test power of 80% for references 104 and 105. To account for the possible non-parametric distribution of the data, 15% more subjects should be added to each group. Another 25% will be added to account for possible dropouts, resulting in 13 participants per group and for greater safety and reliability, 15 patients were established in each group. G*Power 3.1.9.6 was used to perform the calculations.

Materials used in the study:

The biomaterial chosen for this research is the Plenum® OSShp and Plenum® Guide (Brazil) allograft. They are completely synthetic bone grafts and resorbable regenerating membranes (free of animal and human origin).

Plenum® OSShp is a porous synthetic biphasic bioceramic (hydroxyapatite: β - tricalcium phosphate, HA: β-TCP - 70:30%), and the granules are 500 - 1000 µm.

Plenum® Guide is a polydioxanone (PDO)-based synthetic membrane material whose surface morphology closely mimics the extracellular matrix.

Randomization:

All participants will be invited to participate in the research and after signing the informed consent will be randomized into blocks of 4; 60 participants will be randomly divided into 4 groups n=15 Exo (extraction), Exo+Laser (extraction and treatment with 808 nm laser), Exo+Biomat (extraction with biomaterial graft), Exo+Biomat+Laser (extraction and grafting of biomaterial and 808 nm laser treatment). Participants will be randomly allocated by a computer-generated list (Excel) 4.7 CLINICAL PROCEDURE: At the pre-surgical moment, the patient will be submitted to a CT scan (Figure 12) and intraoral scanning (Figure 13) for initial measurement of the vertical and horizontal bone dimensions of the alveolus and between the adjacent teeth of the tooth to be extracted in position in the alveolus and dental arch, and surgical planning, as recommended by the best current dentistry practices, and will sign the Image Use Authorization Term (ANNEX 4). Pre-surgical guidance and delivery of prescriptions with the established drug protocol will also be carried out. All research patients will receive the same post-surgical guidance care (ANNEX 3) and the drug protocol performed for all tooth removal surgery with or without grafting with biomaterials. The tooth will be extracted using an odontosection technique to remove the roots with the least possible trauma. It will not be necessary to lift the soft tissue flap due to the properties of the membrane that will be used, reducing tissue trauma and helping to repair the surgical site. After the extraction, the biomaterial will be added and accommodated to the socket with instruments that allow this insertion and covered by a membrane that will serve as a mechanical barrier, preventing the invagination of the gingival tissue and the formation of keratinized tissue to close the surgical wound so as not to compromise the osseointegration of the bone biomaterial. grafted.

The Exo+Laser and Exo+Biomat+Laser groups will receive, in addition to the drug protocol and guidelines, laser treatment. The Exo and Exo+Biomat groups will use a similar laser device, however, it will not emit irradiation.

In the postoperative period at 3 and 6 months, new intraoral digital scanning and digital computed tomography exams will be performed to take images and perform volumetric analysis with specific software.

ELIGIBILITY:
Inclusion Criteria:

* All genders, aged between 8 and 17 years, without comorbidities, present satisfactory oral hygiene and present a condition of loss of first or second permanent molars

Exclusion Criteria:

* Habitual use of analgesic and anti-inflammatory medication for other comorbidities, present allergies to the proposed drug protocol, in neurological/psychiatric treatment, presence of teeth with lesions to be treated in the same hemiarch of the tooth to be removed, current smoking habit, pregnant or breast-feeding, presenting photosensitivity disorders, with the presence of neoplasia in the oral region; and patients with operative complications whose surgical time exceeds 90 minutes

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Surgical intervention phase | Baseline, pre surgical, 3 and 6 months
  The computed tomography examination will be carried out pre-surgery, with the tooth before extraction and after 3 and 6 months after surgery and the measurements chosen for the dimensional measurement of the alveolar process will refer to the buccolingual thickness of the alveolus. In the orthoradial cut, the limits of the alveolus will be delimited based on the tooth apex to the maximum height of the bone crests. In the most central position, the vertical measurement will be taken and 3 buccolingual cuts will be made, proportional to each other according to the measured vertical measurement; and in each apical, middle and cervical third, measurements will be taken regarding the horizontal dimensions of the alveolus. In the intraoral scanning examination, the mesio-distal measurements will be measured from the mesial bone crest to the distal bone crest, and the buccal-lingual measurements in the most central portion of the dental socket.

SECONDARY OUTCOMES:
Interdental distance | Baseline, pre surgical, 3 and 6 months
  In computed tomography and intraoral scanning, the horizontal distance will be measured with the limit at the mesial and distal bone crest of the alveolus preoperatively with the tooth still in place, 3 and 6 months after extraction, to verify maintenance of the interdental space.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Dalapria, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

REFERENCES:
- [Result] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Result] Petersen PE. The World Oral Health Report 2003: continuous improvement of oral health in the 21st century--the approach of the WHO Global Oral Health Programme. Community Dent Oral Epidemiol. 2003 Dec;31 Suppl 1:3-23. doi: 10.1046/j..2003.com122.x. PMID 15015736
- [Result] De Marchi RJ, Hugo FN, Hilgert JB, Padilha DM. Association between oral health status and nutritional status in south Brazilian independent-living older people. Nutrition. 2008 Jun;24(6):546-53. doi: 10.1016/j.nut.2008.01.054. PMID 18455655
- [Result] Rezaie M, Ghapanchi J, Haghnegahdar A, Khojastehpour L, Khorshidi H, Heidari H. A Radiographic Evaluation of Missing of Permanent First Molars in a Group of Iranian Children and Adults: A Retrospective Study. Int J Dent. 2018 Apr 1;2018:5253965. doi: 10.1155/2018/5253965. eCollection 2018. PMID 29808093
- [Result] Saber AM, Altoukhi DH, Horaib MF, El-Housseiny AA, Alamoudi NM, Sabbagh HJ. Consequences of early extraction of compromised first permanent molar: a systematic review. BMC Oral Health. 2018 Apr 5;18(1):59. doi: 10.1186/s12903-018-0516-4. PMID 29622000
- [Result] Alkhadra T. A Systematic Review of the Consequences of Early Extraction of First Permanent First Molar in Different Mixed Dentition Stages. J Int Soc Prev Community Dent. 2017 Sep-Oct;7(5):223-226. doi: 10.4103/jispcd.JISPCD_222_17. Epub 2017 Sep 18. PMID 29026692
- [Result] Chappuis V, Araujo MG, Buser D. Clinical relevance of dimensional bone and soft tissue alterations post-extraction in esthetic sites. Periodontol 2000. 2017 Feb;73(1):73-83. doi: 10.1111/prd.12167. PMID 28000281
- [Result] Barone A, Aldini NN, Fini M, Giardino R, Calvo Guirado JL, Covani U. Xenograft versus extraction alone for ridge preservation after tooth removal: a clinical and histomorphometric study. J Periodontol. 2008 Aug;79(8):1370-7. doi: 10.1902/jop.2008.070628. PMID 18672985
- [Result] Araujo MG, Lindhe J. Ridge preservation with the use of Bio-Oss collagen: A 6-month study in the dog. Clin Oral Implants Res. 2009 May;20(5):433-40. doi: 10.1111/j.1600-0501.2009.01705.x. PMID 19522974
- [Result] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Ridge alterations following implant placement in fresh extraction sockets: an experimental study in the dog. J Clin Periodontol. 2005 Jun;32(6):645-52. doi: 10.1111/j.1600-051X.2005.00726.x. PMID 15882225
- [Result] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Result] Osburn RC. Preservation of the alveolar ridge: a simplified technique for retaining teeth beneath removable appliances. J Indiana State Dent Assoc. 1974 Jan-Feb;53(1):8-11. No abstract available. PMID 4523604
- [Result] PELTIER LF. The use of plaster of Paris to fill defects in bone. Clin Orthop. 1961;21:1-31. No abstract available. PMID 14485018
- [Result] Artzi Z, Nemcovsky CE. The application of deproteinized bovine bone mineral for ridge preservation prior to implantation. Clinical and histological observations in a case report. J Periodontol. 1998 Sep;69(9):1062-7. doi: 10.1902/jop.1998.69.9.1062. PMID 9776036
- [Result] Faour O, Dimitriou R, Cousins CA, Giannoudis PV. The use of bone graft substitutes in large cancellous voids: any specific needs? Injury. 2011 Sep;42 Suppl 2:S87-90. doi: 10.1016/j.injury.2011.06.020. Epub 2011 Jul 2. PMID 21723553
- [Result] Misch CE, Perez HM. Atraumatic extractions: a biomechanical rationale. Dent Today. 2008 Aug;27(8):98, 100-1. PMID 18717405
- [Result] Saito S, Shimizu N. Stimulatory effects of low-power laser irradiation on bone regeneration in midpalatal suture during expansion in the rat. Am J Orthod Dentofacial Orthop. 1997 May;111(5):525-32. doi: 10.1016/s0889-5406(97)70152-5. PMID 9155812
- [Result] LeGeros RZ. Calcium phosphate materials in restorative dentistry: a review. Adv Dent Res. 1988 Aug;2(1):164-80. doi: 10.1177/08959374880020011101. No abstract available. PMID 3073782
- [Result] Salama R, Burwell RD, Dickson IR. Recombined grafts of bone and marrow. The beneficial effect upon osteogenesis of impregnating xenograft (heterograft) bone with autologous red marrow. J Bone Joint Surg Br. 1973 May;55(2):402-17. No abstract available. PMID 4574991
- [Result] Hoexter DL. Bone regeneration graft materials. J Oral Implantol. 2002;28(6):290-4. doi: 10.1563/1548-1336(2002)0282.3.CO;2. PMID 12498538
- [Result] Landsberg CJ. Implementing socket seal surgery as a socket preservation technique for pontic site development: surgical steps revisited--a report of two cases. J Periodontol. 2008 May;79(5):945-54. doi: 10.1902/jop.2008.070298. PMID 18454676
- [Result] Nemcovsky CE, Artzi Z, Moses O. Rotated palatal flap in immediate implant procedures. Clinical evaluation of 26 consecutive cases. Clin Oral Implants Res. 2000 Feb;11(1):83-90. doi: 10.1034/j.1600-0501.2000.011001083.x. PMID 11168198
- [Result] Sclar AG. Strategies for management of single-tooth extraction sites in aesthetic implant therapy. J Oral Maxillofac Surg. 2004 Sep;62(9 Suppl 2):90-105. doi: 10.1016/j.joms.2004.06.041. PMID 15332186
- [Result] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Result] Jung RE, Siegenthaler DW, Hammerle CH. Postextraction tissue management: a soft tissue punch technique. Int J Periodontics Restorative Dent. 2004 Dec;24(6):545-53. PMID 15626317
- [Result] Davies N, Dobner S, Bezuidenhout D, Schmidt C, Beck M, Zisch AH, Zilla P. The dosage dependence of VEGF stimulation on scaffold neovascularisation. Biomaterials. 2008 Sep;29(26):3531-8. doi: 10.1016/j.biomaterials.2008.05.007. Epub 2008 Jun 9. PMID 18541296
- [Result] Araujo MG, Lindhe J. Socket grafting with the use of autologous bone: an experimental study in the dog. Clin Oral Implants Res. 2011 Jan;22(1):9-13. doi: 10.1111/j.1600-0501.2010.01937.x. Epub 2010 Nov 22. PMID 21091539
- [Result] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Result] Holtrop ME, Cox KA, Glowacki J. Cells of the mononuclear phagocytic system resorb implanted bone matrix: a histologic and ultrastructural study. Calcif Tissue Int. 1982 Sep;34(5):488-94. doi: 10.1007/BF02411290. PMID 6817899
- [Result] Chappard D, Guillaume B, Mallet R, Pascaretti-Grizon F, Basle MF, Libouban H. Sinus lift augmentation and beta-TCP: a microCT and histologic analysis on human bone biopsies. Micron. 2010 Jun;41(4):321-6. doi: 10.1016/j.micron.2009.12.005. Epub 2009 Dec 22. PMID 20060730
- [Result] Fickl S, Fischer K, Petersen N, Happe A, Schlee M, Schlagenhauf U, Kebschull M. Dimensional Evaluation of Different Ridge Preservation Techniques: A Randomized Clinical Study. Int J Periodontics Restorative Dent. 2017 May/Jun;37(3):403-410. doi: 10.11607/prd.2629. PMID 28402351
- [Result] Artzi Z, Weinreb M, Givol N, Rohrer MD, Nemcovsky CE, Prasad HS, Tal H. Biomaterial resorption rate and healing site morphology of inorganic bovine bone and beta-tricalcium phosphate in the canine: a 24-month longitudinal histologic study and morphometric analysis. Int J Oral Maxillofac Implants. 2004 May-Jun;19(3):357-68. PMID 15214219
- [Result] Pasqualini D, Cocero N, Castella A, Mela L, Bracco P. Primary and secondary closure of the surgical wound after removal of impacted mandibular third molars: a comparative study. Int J Oral Maxillofac Surg. 2005 Jan;34(1):52-7. doi: 10.1016/j.ijom.2004.01.023. PMID 15617967
- [Result] Wood DL, Hoag PM, Donnenfeld OW, Rosenfeld LD. Alveolar crest reduction following full and partial thickness flaps. J Periodontol. 1972 Mar;43(3):141-4. doi: 10.1902/jop.1972.43.3.141. No abstract available. PMID 4501971
- [Result] Ngeow WC, Lim D. Do Corticosteroids Still Have a Role in the Management of Third Molar Surgery? Adv Ther. 2016 Jul;33(7):1105-39. doi: 10.1007/s12325-016-0357-y. Epub 2016 Jun 10. PMID 27287853
- [Result] Baxendale BR, Vater M, Lavery KM. Dexamethasone reduces pain and swelling following extraction of third molar teeth. Anaesthesia. 1993 Nov;48(11):961-4. doi: 10.1111/j.1365-2044.1993.tb07474.x. PMID 8250191
- [Result] Tavares MG, Machado AP, Motta BG, Borsatto MC, Rosa AL, Xavier SP. Electro-acupuncture efficacy on pain control after mandibular third molar surgery. Braz Dent J. 2007;18(2):158-62. doi: 10.1590/s0103-64402007000200014. PMID 17982558
- [Result] Seymour RA, Hawkesford JE, Weldon M, Brewster D. An evaluation of different ibuprofen preparations in the control of postoperative pain after third molar surgery. Br J Clin Pharmacol. 1991 Jan;31(1):83-7. doi: 10.1111/j.1365-2125.1991.tb03861.x. PMID 2015175
- [Result] Merigo E, Vescovi P, Margalit M, Ricotti E, Stea S, Meleti M, Manfredi M, Fornaini C. Efficacy of LLLT in swelling and pain control after the extraction of lower impacted third molars. Laser Ther. 2015 Mar 31;24(1):39-46. doi: 10.5978/islsm.15-OR-05. PMID 25941424
- [Result] Kathuria V, Dhillon JK, Kalra G. Low Level Laser Therapy: A Panacea for oral maladies. Laser Ther. 2015 Oct 2;24(3):215-23. doi: 10.5978/islsm.15-RA-01. PMID 26557737
- [Result] Pandeshwar P, Roa MD, Das R, Shastry SP, Kaul R, Srinivasreddy MB. Photobiomodulation in oral medicine: a review. J Investig Clin Dent. 2016 May;7(2):114-26. doi: 10.1111/jicd.12148. Epub 2015 Feb 26. PMID 25720555
- [Result] Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR. The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. 2012 Feb;40(2):516-33. doi: 10.1007/s10439-011-0454-7. Epub 2011 Nov 2. PMID 22045511
- [Result] Rola P, Doroszko A, Derkacz A. The Use of Low-Level Energy Laser Radiation in Basic and Clinical Research. Adv Clin Exp Med. 2014 September-October;23(5):835-842. doi: 10.17219/acem/37263. PMID 25491701
- [Result] Karu TI. [Molecular mechanism of the therapeutic effect of low-intensity laser irradiation]. Dokl Akad Nauk SSSR. 1986;291(5):1245-9. No abstract available. Russian. PMID 3542462
- [Result] Basford JR. Low-energy laser therapy: controversies and new research findings. Lasers Surg Med. 1989;9(1):1-5. doi: 10.1002/lsm.1900090103. No abstract available. PMID 2648091
- [Result] Basford JR. Low intensity laser therapy: still not an established clinical tool. Lasers Surg Med. 1995;16(4):331-42. doi: 10.1002/lsm.1900160404. PMID 7651054
- [Result] Nicola JH, Nicola EM. Wavelength, frequency, and color: absolute or relative concepts? J Clin Laser Med Surg. 2002 Dec;20(6):307-11. doi: 10.1089/104454702320901080. PMID 12513916
- [Result] AboElsaad NS, Soory M, Gadalla LM, Ragab LI, Dunne S, Zalata KR, Louca C. Effect of soft laser and bioactive glass on bone regeneration in the treatment of infra-bony defects (a clinical study). Lasers Med Sci. 2009 May;24(3):387-95. doi: 10.1007/s10103-008-0576-9. Epub 2008 Jun 26. PMID 18581160
- [Result] Cavalcanti TM, Almeida-Barros RQ, Catao MH, Feitosa AP, Lins RD. Knowledge of the physical properties and interaction of laser with biological tissue in dentistry. An Bras Dermatol. 2011 Sep-Oct;86(5):955-60. doi: 10.1590/s0365-05962011000500014. English, Portuguese. PMID 22147036
- [Result] Romao MM, Marques MM, Cortes AR, Horliana AC, Moreira MS, Lascala CA. Micro-computed tomography and histomorphometric analysis of human alveolar bone repair induced by laser phototherapy: a pilot study. Int J Oral Maxillofac Surg. 2015 Dec;44(12):1521-8. doi: 10.1016/j.ijom.2015.08.989. Epub 2015 Sep 14. PMID 26381208
- [Result] Huang YY, Chen AC, Carroll JD, Hamblin MR. Biphasic dose response in low level light therapy. Dose Response. 2009 Sep 1;7(4):358-83. doi: 10.2203/dose-response.09-027.Hamblin. PMID 20011653
- [Result] Karu TI, Kolyakov SF. Exact action spectra for cellular responses relevant to phototherapy. Photomed Laser Surg. 2005 Aug;23(4):355-61. doi: 10.1089/pho.2005.23.355. PMID 16144476
- [Result] Casado PL, Duarte ME, Carvalho W, Esmeraldo da Silva L, Barboza EP. Ridge bone maintenance in human after extraction. Implant Dent. 2010 Aug;19(4):314-22. doi: 10.1097/ID.0b013e3181dec322. PMID 20683288
- [Result] Liu X, Lyon R, Meier HT, Thometz J, Haworth ST. Effect of lower-level laser therapy on rabbit tibial fracture. Photomed Laser Surg. 2007 Dec;25(6):487-94. doi: 10.1089/pho.2006.2075. PMID 18158750
- [Result] Renno AC, McDonnell PA, Parizotto NA, Laakso EL. The effects of laser irradiation on osteoblast and osteosarcoma cell proliferation and differentiation in vitro. Photomed Laser Surg. 2007 Aug;25(4):275-80. doi: 10.1089/pho.2007.2055. PMID 17803384
- [Result] Silveira PC, Silva LA, Freitas TP, Latini A, Pinho RA. Effects of low-power laser irradiation (LPLI) at different wavelengths and doses on oxidative stress and fibrogenesis parameters in an animal model of wound healing. Lasers Med Sci. 2011 Jan;26(1):125-31. doi: 10.1007/s10103-010-0839-0. Epub 2010 Sep 24. PMID 20865435
- [Result] Brignardello-Petersen R, Carrasco-Labra A, Araya I, Yanine N, Beyene J, Shah PS. Is adjuvant laser therapy effective for preventing pain, swelling, and trismus after surgical removal of impacted mandibular third molars? A systematic review and meta-analysis. J Oral Maxillofac Surg. 2012 Aug;70(8):1789-801. doi: 10.1016/j.joms.2012.01.008. Epub 2012 Mar 6. PMID 22398186
- [Result] Kornman KS, Robertson PB. Fundamental principles affecting the outcomes of therapy for osseous lesions. Periodontol 2000. 2000 Feb;22:22-43. doi: 10.1034/j.1600-0757.2000.2220103.x. No abstract available. PMID 11276514
- [Result] Pogrel MA, Chen JW, Zhang K. Effects of low-energy gallium-aluminum-arsenide laser irradiation on cultured fibroblasts and keratinocytes. Lasers Surg Med. 1997;20(4):426-32. doi: 10.1002/(sici)1096-9101(1997)20:43.0.co;2-s. PMID 9142682
- [Result] Lirani-Galvao AP, Jorgetti V, da Silva OL. Comparative study of how low-level laser therapy and low-intensity pulsed ultrasound affect bone repair in rats. Photomed Laser Surg. 2006 Dec;24(6):735-40. doi: 10.1089/pho.2006.24.735. PMID 17199474
- [Result] Barbos Pinheiro AL, Limeira Junior Fde A, Marquez Gerbi ME, Pedreira Ramalho LM, Marzola C, Carneiro Ponzi EA, Oliveira Soares A, Bandeira De Carvalho LC, Vieira Lima HC, Oliveira Goncalves T. Effect of 830-nm laser light on the repair of bone defects grafted with inorganic bovine bone and decalcified cortical osseous membrane. J Clin Laser Med Surg. 2003 Dec;21(6):383-8. doi: 10.1089/104454703322650202. PMID 14709224
- [Result] Gerbi ME, Marques AM, Ramalho LM, Ponzi EA, Carvalho CM, Santos Rde C, Oliveira PC, Noia M, Pinheiro AL. Infrared laser light further improves bone healing when associated with bone morphogenic proteins: an in vivo study in a rodent model. Photomed Laser Surg. 2008 Feb;26(1):55-60. doi: 10.1089/pho.2007.2026. PMID 18248162
- [Result] Lopes CB, Pacheco MT, Silveira L Jr, Duarte J, Cangussu MC, Pinheiro AL. The effect of the association of NIR laser therapy BMPs, and guided bone regeneration on tibial fractures treated with wire osteosynthesis: Raman spectroscopy study. J Photochem Photobiol B. 2007 Dec 14;89(2-3):125-30. doi: 10.1016/j.jphotobiol.2007.09.011. Epub 2007 Oct 1. PMID 17981047
- [Result] Rochkind S, Kogan G, Luger EG, Salame K, Karp E, Graif M, Weiss J. Molecular structure of the bony tissue after experimental trauma to the mandibular region followed by laser therapy. Photomed Laser Surg. 2004 Jun;22(3):249-53. doi: 10.1089/1549541041438579. PMID 15315733
- [Result] Coombe AR, Ho CT, Darendeliler MA, Hunter N, Philips JR, Chapple CC, Yum LW. The effects of low level laser irradiation on osteoblastic cells. Clin Orthod Res. 2001 Feb;4(1):3-14. doi: 10.1034/j.1600-0544.2001.040102.x. PMID 11553080
- [Result] Ninomiya T, Miyamoto Y, Ito T, Yamashita A, Wakita M, Nishisaka T. High-intensity pulsed laser irradiation accelerates bone formation in metaphyseal trabecular bone in rat femur. J Bone Miner Metab. 2003;21(2):67-73. doi: 10.1007/s007740300011. PMID 12601569
- [Result] Dalapria V, Marcos RL, Bussadori SK, Anselmo G, Benetti C, da Silva Santana ACA, Marinho NSR, Pinto RS, de Sales RS, de Franca LS, Deana AM. LED photobiomodulation therapy combined with biomaterial as a scaffold promotes better bone quality in the dental alveolus in an experimental extraction model. Lasers Med Sci. 2022 Apr;37(3):1583-1592. doi: 10.1007/s10103-021-03407-w. Epub 2021 Nov 12. PMID 34767116
- [Result] Obradovic RR, Kesic LG, Pesevska S. Influence of low-level laser therapy on biomaterial osseointegration: a mini-review. Lasers Med Sci. 2009 May;24(3):447-51. doi: 10.1007/s10103-008-0573-z. Epub 2008 Jun 20. PMID 18566853
- [Result] Rosero KAV, Sampaio RMF, Deboni MCZ, Correa L, Marques MM, Ferraz EP, da Graca Naclerio-Homem M. Photobiomodulation as an adjunctive therapy for alveolar socket preservation: a preliminary study in humans. Lasers Med Sci. 2020 Oct;35(8):1711-1720. doi: 10.1007/s10103-020-02962-y. Epub 2020 Jan 22. PMID 31970564
- [Result] Araujo MG, da Silva JCC, de Mendonca AF, Lindhe J. Ridge alterations following grafting of fresh extraction sockets in man. A randomized clinical trial. Clin Oral Implants Res. 2015 Apr;26(4):407-412. doi: 10.1111/clr.12366. Epub 2014 Mar 12. PMID 24621203